CLINICAL TRIAL: NCT01774695
Title: An Intervention to Improve Physical Activity in IBS Patients Has Long Term Positive Effects
Brief Title: Physical Activity in IBS - a Long Term Follow up
Acronym: IBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Magnus Simrén, MD, PhD, Sahlgrenska University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VGFOUSA-181101
Record Dates: First submitted 2013-01-08; First posted 2013-01-24 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Irritable Bowel Syndrome (IBS)
Keywords: IBS; physical activity; exercise
MeSH Terms: conditions — Irritable Bowel Syndrome; Motor Activity

ARMS (1):
- Control and intervention (Other): In the first study half of the subjects first served as controls for 12 weeks and then they went through the intervention. The other half only went through the intervention.
  Interventions: Behavioral: Increased physical activity

INTERVENTIONS:
Behavioral: Increased physical activity — The subjects were encouraged to increase their level of physical activity for 12 weeks in the previous study.
  The advice was individual but was based on the recommendations of the Swedish National Institute of health. The recommendation for increasing cardiorespiratory fitness is 20-60 minutes of moderate to vigorous intensive physical activity 3 to 5 days per week.

SUMMARY:
Increased physical activity has in the investigators recent study been shown to improve symptoms in irritable bowel syndrome (IBS). The aim of this study was to assess the long term effects of the investigators previous intervention in IBS patients to improve physical activity. The investigators aimed to assess the long term effects on IBS symptoms as well as quality of life, fatigue, depression and anxiety.

DETAILED DESCRIPTION:
86 patients who had been included in the investigators previous study "Physical Activity Improves Symptoms in Irritable Bowel Syndrome: A Randomized Controlled Trial" were contacted and asked to participate in a long term follow up 5 years after the previous study. The subjects attended one visit at which they underwent a bicycle ergometer test to calculate the oxygen uptake and filled out questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Baseline data from the previous study

Exclusion Criteria:

* pregnancy
* organic gastrointestinal disorders
* cardiac disease
* respiratory disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2011-06; Primary Completion 2011-09 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
IBS Severity Scoring System (IBS-SSS) | Change between baseline and follow up after five years
  The IBS-SSS consists of visual analog scales and is divided into two subscales, an overall IBS score and an extra colonic score. The IBS score contains questions regarding pain severity, pain frequency, abdominal bloating, bowel habit dissatisfaction, and life interference. The extra colonic score contains questions regarding vomiting, gas, belching, satiety, headache, fatigue, musculoskeletal pain, heartburn, dysuria and urgency. Each subscale ranges from 0 to 500, with higher scores meaning more severe symptoms. A reduction of 50 is considered to be adequate to detect a clinical improvement.

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) | Change between baseline and follow up after 5 years
  HADS was developed for medical outpatients and consists of 14 items, each using a 4-graded Likert scale (0-3). The scale is divided into two subscales, anxiety and depression. Each subscale ranges from 0 to 21, where high score means more severe symptoms.
IBS Quality of Life (IBS-QoL) | Change between baseline and follow up after 5 years
  The IBS-QOL is a disease specific instrument measuring HRQOL. It consists of 30 items which measures nine dimensions; emotional functioning, mental health, sleep, energy, physical functioning, diet, social role, physical role and sexual relations. For each subscale the scores are transformed to range from 0 to 100; 100 representing the best possible disease specific quality of life.
Short Form 36 (SF-36) | Change between baseline and follow up after 5 years
  SF-36 was used to assess the general HRQOL. SF-36 includes 36 items which are divided into eight subscales; physical functioning, physical role, body pain, general health perceptions, vitality, social functioning, emotional role and mental health. For each subscale the raw scores are transformed into a scale from 0 to 100, with 100 representing the best possible HRQOL.
Fatigue Impacts Scale(FIS) | Change between baseline and follow up after 5 years
  This scale was initially developed for patients with chronic fatigue syndrome and has previously been used in studies in IBS patients.11 The scale consists of 40 questions divided into three subscales, physical functioning (10 items), cognitive functioning (10 items) and psychosocial functioning (20 items). The subjects are asked to rate to which extent fatigue has caused problems for them during the previous month. Each item consists of a statement and the subject should rate 0 to 4 where 0 means 'no problem' and 4 means 'extreme problem'.

OTHER OUTCOMES:
Oxygen uptake | Change between baseline and at follow up after 5 years
  The oxygen uptake was calculated from a submaximal cycle (Monark Ergomedic 839). ergometer test according to Astrand.

CONTACTS AND LOCATIONS:
Locations (1):
- Dept of Internal Medicine, Sahlgrenska University Hospital, Gothenburg, Sweden

REFERENCES:
- [Background] Johannesson E, Simren M, Strid H, Bajor A, Sadik R. Physical activity improves symptoms in irritable bowel syndrome: a randomized controlled trial. Am J Gastroenterol. 2011 May;106(5):915-22. doi: 10.1038/ajg.2010.480. Epub 2011 Jan 4. PMID 21206488